CLINICAL TRIAL: NCT00537368
Title: A Phase 1 Study of CNTO 888, a Human Monoclonal Antibody Against CC-Chemokine Ligand 2 in Subjects With Solid Tumors
Brief Title: First Study of the Safety of CNTO 888 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013699
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Cancer
Keywords: infusion; CNTO 888; Phase 1; solid tumor; cancer
MeSH Terms: conditions — Neoplasms | interventions — carlumab

INTERVENTIONS:
Drug: CNTO 888

SUMMARY:
The purpose of this study is to determine if CNTO 888 is safe and to determine how long CNTO 888 stays in the body and what effects it might have on cancer tumors.

DETAILED DESCRIPTION:
CNTO 888 is a monoclonal antibody. Antibodies are substances in the body that are involved in many biological processes. CNTO 888 is thought to work by blocking a protein called CC-Chemokine Ligand 2 (CCL2). In research studies CCL2 has been shown to increase the growth of new blood vessels which help the tumor to survive. When new blood vessels do not grow, tumors cannot get the food or oxygen they need to grow. Blocking CCL2 may help fight disease.This study consists of two parts, Part A and Part B. In Part A, five different groups of patients will be treated with five different, increasing dose levels of CNTO 888. In Part B, two of the dose levels of CNTO 888 will be tested further in different treatment schedules. CNTO 888 is given by intravenous (into the vein) infusion. Between 1 and 30 patients with advanced cancer will take part in Part A of the study. Between 24 and 33 patients with advanced cancer will take part in Part B of the study.There are three phases in part A of the study. Screening phase, which may last up to 4 weeks. Treatment phase, which may last up to 8 weeks (4 treatments) and can be extended for an extra 9 weeks (4 extra treatments) in case the patient's tumor is not getting bigger. The total treatment period could be up to 17 weeks. Follow up phase will include an end of treatment visit 4 weeks after the last infusion of CNTO 888, visits through week 18 after last infusion as well as long term collection of follow up data. After Part A is completed, up to two doses will be selected for evaluation in part B. In Part B, patients will be placed into one of 3 study groups. There are three phases in Part B of this study. The screening phase, which may last up to 4 weeks. The treatment phase, which may last up to 9 weeks (4 treatments). If the patient's tumor is not getting bigger, the patient's treatment phase may be extended up to 12 weeks (4 treatments). The total treatment period could be up to 21 weeks. The follow up phase will include an end of treatment visit 4 weeks after the last infusion of CNTO 888, visits through week 18 after last infusion as well as long-term collection of follow up data. Safety and effectiveness evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and collection of information about the occurrence and severity of adverse events. In Part A of this study, patients will receive either 0.3 , 1.0, 3.0, 10, or 15 mg/kg CNTO 888. The time between the first and second infusion is 4 weeks, with all of the following infusions will be given 2 weeks apart. Patients eligible for Part B will be assigned to either the lower dose selected from Part A, given every 2 weeks or the higher dose selected from Part A given either every 2 weeks or every 3 weeks. All patients may be in the study for 18 weeks after their last infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumors that have progressed on or after all available standard therapy
* Histological or cytological documentation of specific tumor type
* Evidence of measurable or evaluable metastatic disease
* Anticipated life expectancy is >= 12 weeks

Exclusion Criteria:

* Treatment with systemic cancer therapy or local radiotherapy within 4 weeks
* Received any investigational drug/agent within 4 weeks
* Major surgery within 4 weeks of first dose of study agent
* Serious concurrent illness (medical or psychiatric), altered mental status (eg, dementia) or any uncontrolled medical condition (eg, uncontrolled diabetes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-09; Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and pharmacokinetics (rate of movement in the body and then the clearance) of CNTO 888 administered as multiple intravenous (IV) infusions in patients with solid tumors throughout the course of the study.

SECONDARY OUTCOMES:
Assess the pharmacodynamics (action of drug on body systems), immune response and clinical effects (tumor response and time to disease progression) of CNTO888 when administered as multiple IV infusions in patients with solid tumors throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.